CLINICAL TRIAL: NCT03120767
Title: Wellness Initiative at New York University
Acronym: WIN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to inability to enroll patients
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-02124
Record Dates: First submitted 2017-03-24; First posted 2017-04-19 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Health Promotion
MeSH Terms: interventions — Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Condition 1 (Experimental): enrolled in the Risk and Resilience course during Fall 2017 and directly encouraged to participate in the Founders Living and Learning Community wellness activities for the Fall of 2017 (Coordinated Wellness Programming)
  Interventions: Behavioral: Risk and Resilience; Behavioral: Coordinated Wellness Programming
- Condition 2 (Active Comparator): enrolled in the Risk and Resilience course in Spring 2018, and not directly encouraged to participate in the WIN Living and Learning Community wellness activities
  Interventions: Behavioral: Risk and Resilience
- Condition 3 (No Intervention): a control group that receives none of the interventions during the first year. This group will instead receive an online pamphlet that contains a number of wellness tips and advice for first-year students. Condition 3 participants have access to the WIN Living and Learning Community wellness activities in Fall of 2017 and Spring of 2018, but are not directly encouraged to participate.

INTERVENTIONS:
Behavioral: Risk and Resilience — The "Risk and Resilience" course is a 14-week undergraduate seminar that is grounded in the current understanding of adolescent and young adult development, neuroscience, and positive psychology. Students will learn about key areas proven to enhance wellness, including communication, executive functioning, social support, self-efficacy, emotion regulation, and sense of purpose. Students will learn about healthy exercise, nutrition, and sleep habits, and develop skills in core components of cognitive-behavior therapy, mindfulness, and organizational skills.
  Arms: Condition 1; Condition 2
Behavioral: Coordinated Wellness Programming — During the Fall of 2017, wellness activities will be provided within Founders Hall that support the theories and skills being taught in the "Risk and Resilience" course occurring in the same semester.
  Arms: Condition 1

SUMMARY:
The goal of this study is to evaluate the effect on first-year college students of participation in a 14-week seminar course and residential housing wellness activities.

DETAILED DESCRIPTION:
WIN has been designed to enhance student wellness and personal success during college and after graduation from New York University. The program is grounded in the current understanding of adolescent and young adult development, neuroscience, and positive psychology and aims to increase resilience within students by building knowledge and skills in key areas proven to enhance wellness, including communication, executive functioning, social support, cognitive behavioral techniques, stress management, emotion regulation, and sense of purpose. WIN will achieve these aims by teaching this knowledge and skills to students in a class ("Risk and Resilience") and via participation in various activities within a residential Living and Learning Community. Students will not only receive training and support in establishing healthy exercise, nutrition, and sleep habits, students will also be taught core components of cognitive-behavior therapy, mindfulness, and organizational skills training.

In tandem with the implementation of WIN,the effectiveness of the program will be evaluated. A research study will offer benefits: first, it will provide the college with data for future estimations of student interest to assist in further expanding the scope of wellness; and second, it will provide the Child Study Center at NYU with the opportunity to explore the impact of teaching resilience skills to first-year college students and to modify, if appropriate course content to improve effectiveness.

A longitudinal study at NYU beginning in Fall of 2017 of 175 first-year students, who are randomly assigned to one of three conditions after consenting to participate in the research.

200 participants will be recruited during Spring and Summer of 2017 from the incoming first-year students who will begin classes in Fall 2017. It is anticipated that of the 200 enrolled via electronic assent prior to the beginning of the fall 2017 semester, some may not attend NYU and some may rethink the decision to participate and then not follow up with providing informed consent. As such, there will be over-enrolling via preliminary electronic assent so that the following enrollment can be achieved:

175 students will be assigned randomly into one of three conditions:

* 50 students to Condition 1 (enrolled in the Risk and Resilience course during Fall 2017 and directly encouraged to participate in the Founders Living and Learning Community wellness activities for the Fall of 2017)
* 75 students to Condition 2 (waitlisted to be enrolled in the Rick and Resilience course until Spring 2018, and not directly encouraged to participate in the WIN Living and Learning Community wellness activities)
* 50 students to Condition 3 (a control group that receives none of the interventions during the first year). This group will instead receive an online pamphlet that contains a number of wellness tips and advice for first-year students. Participants have access to the WIN Living and Learning Community wellness activities in Fall of 2017 and Spring of 2018, but are not directly encouraged to participate.

The progress of these 175 students will be measured at frequent intervals throughout the first and subsequent years at college, beginning with a baseline assessment battery once participants provide written informed consent in Fall of 2017, followed by a second survey in Winter 2018, another survey at the end of the academic year (May 2018), and then annually thereafter. In addition to collecting demographic factors (age, gender, race, ethnicity, and relationship status), the study will utilize empirically-based measures that will be self-reported by the students, using an online survey tool. These measures will capture a series of attributes that have been demonstrated as being important factors in psychological well-being, including:

* Perceived stress
* Depressive symptoms
* Anxiety symptoms
* Dysfunctional attitudes
* Risk behaviors (smoking, sexual activity, alcohol and drug usage, etc.)
* Coping skills
* Interpersonal communication
* Use of Cognitive-Behavioral Therapy techniques
* Health behaviors (exercise, nutrition, sleep, etc.)

Additional data will be collected to measure academic achievement, such as grade-point average and persistence in college.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* a student at NYU (Ascertained by their nyu.edu email address)
* residing in Founder's Hall (corroborated by NYU Housing)

Exclusion Criteria:

* Provided the potential participant has met the above inclusion criteria, there are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | Change from Baseline to Immediate Post 5 months later; Change from Immediate Post to Follow-Ups (Follow-Ups begin 4 months after Post and continue annually for up to the next 36 months)
  measures subjective experience of stress

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale | Change from Baseline to Immediate Post 5 months later; Change from Immediate Post to Follow-Ups (Follow-Ups begin 4 months after Post and continue annually for up to the next 36 months))
  Measures clinically significant depressive symptomatology
Beck Anxiety Inventory | Change from Baseline to Immediate Post 5 months later; Change from Immediate Post to Follow-Ups (Follow-Ups begin 4 months after Post and continue annually for up to the next 36 months)
  Measures clinically significant anxious symptomatology
Dysfunctional Attitudes Scale | Change from Baseline to Immediate Post 5 months later; Change from Immediate Post to Follow-Ups (Follow-Ups begin 4 months after Post and continue annually for up to the next 36 months)
  Measures to what extent respondents hold attitudes or beliefs that hinder performance
American College Health Association-National College Health Assessment II | Change from Baseline to Immediate Post 5 months later; Change from Immediate Post to Follow-Ups (Follow-Ups begin 4 months after Post and continue annually for up to the next 36 months)
  a national college survey that asks about a variety of college student behaviors, such as risk-taking behaviors, alcohol consumption, nutrition, etc.
Brief Cope | Change from Baseline to Immediate Post 5 months later; Change from Immediate Post to Follow-Ups (Follow-Ups begin 4 months after Post and continue annually for up to the next 36 months)
  measures methods by which respondents cope with stressors in their lives
Interpersonal Communication Skills Inventory | Change from Baseline to Immediate Post 5 months later; Change from Immediate Post to Follow-Ups (Follow-Ups begin 4 months after Post and continue annually for up to the next 36 months)
  measures interpersonal components of effective communication: an adequate self-concept; the ability to be a good listener; the skills of expressing one's thoughts and ideas clearly; being able to cope with emotions; and the willingness of disclose oneself to others
Cognitive-Behavioral Therapy Skills Questionnaire | Change from Baseline to Immediate Post 5 months later; Change from Immediate Post to Follow-Ups (Follow-Ups begin 4 months after Post and continue annually for up to the next 36 months)
  measures use of Cognitive-Behavioral Therapy techniques: behavioral activation and cognitive restructuring

CONTACTS AND LOCATIONS:
Overall Officials: Jess Shatkin, MD, MPH, Principal Investigator — New York University

IPD SHARING:
Plan to Share IPD: No